CLINICAL TRIAL: NCT07057687
Title: Investigation of Short- and Long-Term Effects of Mulligan Mobilization Technique and Relaxation Technique Applied to Patients With Non-Specific Chronic Low Back Pain: A Single-Blind, Randomized Controlled Study
Brief Title: Non-Specific Chronic Low Back Pain Treatment Methods
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Pınar ATAK ÇAKIR, assistant professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-5282
Record Dates: First submitted 2025-06-27; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Non-Specific Chronic Low Back Pain
Keywords: Pain; Relaxation; Chronic Low Back Pain; Mobilization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mulligan Treatment Group (Experimental): Application of the Technique: The direction of the technique will be shaped according to the direction of movement of the patient's pain. If the patient's pain occurs during flexion, flexion will be applied, if it occurs during extension, extension SNAGS will be applied. In the flexion SNAGS application, the physiotherapist places the mobilization belt at the patient's spina iliaca anterior superior (SIAS) level while the patient is sitting or standing. The physiotherapist places his hand, thumbs or the hypothenar part of the hand parallel to the spinous processes one level above the relevant segment. Then, he asks the patient to flex until he feels pain. The physiotherapist continues the flexion by applying force towards the cranium with his hand. After waiting for a while at the end point, the starting position is returned. During this time, the physiotherapist maintains the natural shift in the facet joint. If the pain does not disappear, the application is applied unilaterally.
  Interventions: Other: Mulligan Treatment Group
- Relaxation Techniques Group (Experimental): The individual will be in a sitting or lying position without muscle tension, and progressive relaxation will be provided with verbal commands given for each body part in order. The patient is asked to place their hand on their abdomen and by applying light resistance, they are provided with the direction in which the breath will go. During diaphragmatic breathing, the person breathes deeply and slowly through the nose and out through the mouth for 5-7 seconds, holds it for 2 seconds and exhales for 6-8 seconds. During this time, the abdomen is inflated in 4 directions and care is taken to ensure that there is no auxiliary muscle activity. First, after taking a deep breath, the muscles are tensed, this tension is maintained for 5-7 seconds and then the muscles are relaxed (8-10 seconds). This application will be applied in 3 sets, with 5/6 repetitions and then returning to calm/normal breathing. The treatment will be applied 3 days a week and will last for 4 weeks.
  Interventions: Other: Relaxation Techniques Group
- Conventional Physical Therapy Group (Active Comparator): Conventional physical therapy applied to patients consists of Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound (US) and Hot Pack. TENS will be applied for 20 minutes at a frequency of 100 hertz. US will be applied for 5 minutes at an intensity of 1.2-1.5 W/cm2. Hot Pack will be applied for 20 minutes. Treatment will be applied to the lumbar region. Application will be made 3 days a week for 4 weeks.
  Interventions: Other: Conventional Physical Therapy Group

INTERVENTIONS:
Other: Conventional Physical Therapy Group — Conventional physical therapy applied to patients consists of Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound (US) and Hot Pack. TENS will be applied for 20 minutes at a frequency of 100 hertz. US will be applied for 5 minutes at an intensity of 1.2-1.5 W/cm2. Hot Pack will be applied for 20 minutes. Treatment will be applied to the lumbar region. Application will be made 3 days a week for 4 weeks.
  Arms: Conventional Physical Therapy Group
Other: Relaxation Techniques Group — The individual will be in a sitting or lying position without muscle tension, and progressive relaxation will be provided with verbal commands given for each body part in order. The patient is asked to place their hand on their abdomen and by applying light resistance, they are provided with the direction in which the breath will go. During diaphragmatic breathing, the person breathes deeply and slowly through the nose and out through the mouth for 5-7 seconds, holds it for 2 seconds and exhales for 6-8 seconds. During this time, the abdomen is inflated in 4 directions and care is taken to ensure that there is no auxiliary muscle activity. First, after taking a deep breath, the muscles are tensed, this tension is maintained for 5-7 seconds and then the muscles are relaxed (8-10 seconds). This application will be applied in 3 sets, with 5/6 repetitions and then returning to calm/normal breathing. The treatment will be applied 3 days a week and will last for 4 weeks.
  Arms: Relaxation Techniques Group
Other: Mulligan Treatment Group — Application of the Technique: The direction of the technique will be shaped according to the direction of movement of the patient's pain. If the patient's pain occurs during flexion, flexion will be applied, if it occurs during extension, extension SNAGS will be applied. In the flexion SNAGS application, the physiotherapist places the mobilization belt at the patient's spina iliaca anterior superior (SIAS) level while the patient is sitting or standing. The physiotherapist places his hand, thumbs or the hypothenar part of the hand parallel to the spinous processes one level above the relevant segment. Then, he asks the patient to flex until he feels pain. The physiotherapist continues the flexion by applying force towards the cranium with his hand. After waiting for a while at the end point, the starting position is returned. During this time, the physiotherapist maintains the natural shift in the facet joint. If the pain does not disappear, the application is applied unilaterally.
  Arms: Mulligan Treatment Group

SUMMARY:
In Turkish society, almost all people experience back pain. When this pain lasts longer than 3 months and is not related to any cause, it is called "non-specific chronic back pain". The source of back pain is often not known for sure. While it can be seen with some physical loads; since humans are biopsychosocial beings, it is possible to say that psychological factors can also cause this pain. Along with the pain, the quality of life and functionality of people are negatively affected. In order to avoid situations such as loss of work, loss of muscle strength or depression, treatment should be at the center of the individual and a multidisciplinary health team. Many treatment methods are used for back pain, these are pharmacological and non-pharmacological methods. One of the non-pharmacological methods is physical therapy. Physiotherapy methods also have many contents such as mobilization, relaxation, massage, electrotherapy. The physiotherapy methods to be used within the scope of this research include conventional treatment (TENS, US and Hot Pack) application. The Mulligan mobilization technique (Continuous Natural Apophyseal Gliding technique, which is the same as the natural gliding movement of the vertebrae) involves manual application. The relaxation technique involves deep-slow diaphragmatic breathing and the application of progressive relaxation exercise with verbal commands. Individuals between the ages of 18-60 who have been diagnosed with back pain that has not been caused by any reason and has lasted longer than 3 months will be included in the study. The study is planned to be conducted with 45 participants and they will be asked to fill out a "voluntary consent form" before participation. The study consists of 3 groups: conventional (control) group, mobilization group and relaxation group. Conventional treatment will be applied to each group and mobilization and relaxation techniques will be applied in addition to the group determined as a result of randomization. The treatment lasts 4 weeks in certain protocols. 3 evaluations will be made at the beginning, end and 3 months after the treatments. Demographic information, pain and perception questionnaires, shortness test, mobility test, quality of life questionnaire and joint range of motion measurement will be used within the scope of the evaluation.

DETAILED DESCRIPTION:
Considering today's living conditions, people are likely to experience pain in their bodies. One of the most common places where pain occurs is the lumbar region. Low back pain is the leading cause of disability worldwide and has the highest prevalence among musculoskeletal disorders. Many people experience low back pain at least once in their lives. In most cases of acute low back pain, the symptoms disappear and heal on their own. However, in some people, the symptoms persist and this condition can turn into chronic pain. (1) If this low back pain lasts longer than 12 weeks without any neurological findings or obvious structural pathology, it is called Non-Specific Chronic Low Back Pain (NSCLBP). Chronic low back pain can occur at any age and gender. The prognosis is usually not good and significantly affects the patient's daily life activities as well as work performance. (2) Low back pain has many etiologies and is a multifactorial disease, meaning that it is very important to analyze risk factors correctly. (3) Careful evaluation of the factors causing low back pain will be especially important in determining the treatment approach. Many conditions such as incorrect posture while working or sitting in daily life, sedentary lifestyle and inadequate physical activity, overweight and obesity, heavy loads, psychosocial influences, frequent weight lifting or various traumas are among the risk factors affecting low back pain. Some psychological or genetic/hormonal diseases, fractures and postural deformities have also been associated with low back pain secondarily. (2) As in all diseases, evaluation is also very important in NSKBA. A good evaluation will bring the right treatment, and the right treatment will bring recovery. Before the evaluation, the patients' gender, age, body mass index, marital status and who they live with, educational status, previous or ongoing diseases, existing habits such as smoking, occupational status, and all personal information should be learned together with the existence of factors that may affect them and their socioeconomic characteristics. (4) As a result of personal information, it is possible to comment on the source of back pain in some cases, but obtaining definite information from the patient about when and how the pain started will provide a healthier approach. The patient who receives appropriate medical treatment, physical therapy and even surgical treatment when necessary, will have pain relief and tissue healing will occur within a certain period of time. In cases where this healing does not occur, some negative events will develop. Long-lasting pain creates distress, anxiety, depression and reluctance. Since the patient does not want to move due to pain and has limitations, their condition and resistance decrease. This situation brings with it a life dependent on others, the patient develops self-doubt and develops a behavioral model dependent on the people around them, those who provide their medical care and drugs. (5) In this respect, treatment should be carried out carefully together with the patient, his/her relatives and a multidisciplinary team.

Correct assessment and treatment of chronic pain requires a harmonious team effort. The goals we try to achieve in treatment are: Controlling and reducing pain, increasing functional physical activities, reducing disability, eliminating distress and anxiety, regulating and reducing sickness behavior, reducing chronic inefficiency and educating the patient. The basic principle in chronic low back pain is multidisciplinary treatment. Both pharmacological and non-pharmacological methods are applied in the treatment of NSKBA. (5) The aim of medical (pharmacological) treatment is to alleviate symptoms, i.e. it does not eliminate the source of pain. Exercise therapy, psychological treatment, weight control or professional arrangements are also important. In addition to medical treatment, the patient should make functional exercise a lifestyle and should regulate their medications as they are used regularly and add them to their daily routine. Another treatment method is non-pharmacological complementary treatment methods, which include approaches such as exercise, yoga, ozone, hydrotherapy, meditation, reflexology, homeopathy, prolotherapy, aromatherapy, lumbar corset, physical therapy modalities, manipulation, mobilization, massage, acupuncture, behavioral treatment, back schools. (2)(3) Mulligan mobilization techniques (MMT), one of the treatment methods, have gained increasing popularity in the treatment of low back pain in recent years. (6) This technique, developed by Brian Mulligan in the 1980s, includes NAGS (Natural Apophyseal Shift), SNAGS (Continuous Natural Apophyseal Shift) and MWM (Mobility with Movement) applications. (7) The aim of MMT is to correct the biomechanical disorder in the joint. (8) An important spine technique within the Mulligan mobilization concept is continuous natural apophyseal shift (SNAGS) (6). SNAGS are accessory glides performed simultaneously with active movement in a painful or limited range of motion. (7) The glide direction is along the plane of the facet joints and in the weight-bearing position. (9) The shape and direction of the glide varies according to the spinal level segment to be applied. (8) During the application, there should be no pain other than palpation and pressure pain. If pain occurs other than these conditions, mobilization is stopped. If there is no decrease in complaints while the technique is applied, the application should not be insisted on and other treatment methods should be tried. (9) In a 2018 review, Mulligan Mobilization Techniques were found to provide medium and short-term effects on pain and disability in patients with low back pain (10); however, it was stated in the review that the long-term follow-up of the effectiveness of mobilization could not be investigated. In a study conducted in our country in 2022, it was possible to monitor the long-term results of many outcome measures without any deficiencies in the groups. In the real MMT group, changes began to be seen in many parameters at the end of the five-week treatment and the effect of mobilization could be maintained for a long period of six months. Special improvements were observed in the disability and functionality parameters in the 3rd and 6th months compared to the 5th week, and significant changes were detected in these parameters between the groups. (11) Another method that can be applied in the treatment includes relaxation techniques. People use various relaxation techniques to cope with pain. These methods; breathing exercises, massage, walking/exercise, yoga, meditation, autogenic training, biofeedback, laughter therapy, hypnosis, progressive muscle relaxation, listening to music, taking a shower, sleeping, using herbal teas, practicing positive thinking, chatting and distracting others. (12)(13)(14) These types of techniques create cognitive awareness in physiological and psychological contexts, control stress and provide nervous system regulation, and also increase the pain threshold and increase resistance to pain. (12) In order to use relaxation techniques, the individual must be in a calm environment, in a comfortable position and focused. The most commonly used relaxation technique is deep and slow diaphragmatic breathing exercise. For diaphragmatic breathing, the individual sits or lies down without muscle tension and breathes in through the nose and out through the mouth. During this time, the abdomen is inflated in 4 directions and care is taken to ensure that there is no auxiliary muscle activity. (15) One of the techniques applied in combination with breathing exercises, Jacobson progressive relaxation exercise is defined as "a method that provides relaxation throughout the body by voluntary and regular relaxation of large muscle groups in the human body". (16) Jacobson progressive relaxation technique creates a feeling of increasing relaxation with commands. This technique basically involves contracting and relaxing muscles or muscle groups in order, and is also called "sequential muscle relaxation technique". The basis of progressive relaxation is to contract the determined muscles while inhaling and to relax these muscles while exhaling. (17)(18) Jacobson states that in the presence of complete relaxation including peripheral body parts, the emotional states of individuals will not be negatively affected and physical relaxation will also bring mental relaxation. In the literature, it has been determined that this technique provides significant improvement in health problems such as tension-type headache, stress, low back pain, hypertension, anxiety, chronic tinnitus, decreased sleep quality, immune deficiencies of the elderly, and undesirable effects of chemotherapy. There is no sufficient content created for its long-term effectiveness in chronic low back pain and its comparison with any mechanical application. During the application of progressive relaxation exercise, all body muscles such as arms, neck, shoulder, chest, abdomen, thighs, legs, feet and fingers are used, including both body parts. First, it is applied by taking a deep breath, then tensing the determined muscles for 5-7 seconds, then maintaining this tension and then relaxing the muscles. (16) Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound (US) and thermal agents (hotpack-coldpack), which are the most frequently applied physical therapy modalities to patients with chronic low back pain, constitute the content of conservative treatment. In a meta-analysis examining the effectiveness of these conservative treatments, it was reported that there was strong evidence for the short-term effectiveness of exercise in particular and it was observed that there was no significant difference in terms of recovery in the conservative treatment group. (19) The goals we want to achieve as a result of this research are to provide guidance on how to approach individuals in the treatment of chronic low back pain. The differences that may occur between the treatment groups will provide us with information on whether the source of the pain is physical or psychological, in other words, it will be an answer to the question of whether these patients need mobility of the spine or relaxation of the body. In addition, we will examine the long-term effectiveness of the treatments and determine which treatment approach is more effective in providing permanence. It has been proven by studies that conventional treatment alone will not be sufficient, and we aim to observe how effective the two methods that are widely used are. As a result of the evaluations, we aim to observe an increase in functionality compared to the beginning, a change in pain perception, an increase in joint range of motion, and an increase in the quality of life of individuals. The possibility that both methods will provide positive results at different rates will provide us with the opportunity to compare the superiority of the methods used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Non-specific low back pain lasting at least 12 weeks
2. Pain must be at least 3 and at most 7 on the Visual Analog Scale (VAS)
3. Age range 18-60
4. Diagnosed by a physician

Exclusion Criteria:

1. Fractures in the spine
2. Pregnancy
3. Cardiac and/or pulmonary diseases
4. Deformities in the spine
5. Surgery in the spine within the last year
6. Systemic diseases
7. Advanced osteoporosis
8. Disc herniation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Recorded 8 weeks and 3 months after the end of treatment
  Pain intensity will be measured according to VAS. The scale consists of a 10 cm line. There are numbers from 0 to 10 on this line. It will be explained to the patient that 0 means no pain and 10 is the last point of unbearable pain. The patient will be asked to mark the level that is most suitable for him/her on this scale.

SECONDARY OUTCOMES:
McGill Melzack Pain Questionnaire | Recorded 8 weeks and 3 months after the end of treatment
  The survey, first developed by Melzack and Katz in 1971, received its Turkish version in 2003. The survey consists of four sections. In the first section, the patient marks the body part or parts affected by the pain. If the pain is coming from deep inside, the patient is asked to indicate it with the letter 'D' and if it is on the body surface, the patient is asked to indicate it with the letter 'Y'. In the second section, the patient is asked what their pain is like. There are 20 word groups that include words that define pain in terms of sensory, perception and evaluation. The patient marks the words they find appropriate from the appropriate group. One appropriate word can be marked from each group, and if none of them are appropriate, the entire word group can be skipped. In the third section, the relationship between pain and time is asked, and what decreases or increases pain is also asked. In the fourth section, the patient is asked questions to determine the severity of pain.
Goniometric Measurement | Recorded 8 weeks and 3 months after the end of treatment
  Flexion and extension measurements are made with the patient standing, the pivot point of the goniometer is placed on the lateral trunk projection of the lumbosacral joint. The fixed arm is placed on the lateral midline of the femur, and the mobile arm is placed parallel to the lateral trunk midline towards the axilla. The patient will then be asked to perform active flexion/extension.
Hand-Ground Distance Measurement | Recorded 8 weeks and 3 months after the end of treatment
  When measuring the hand-to-ground distance, the patient stands with the feet parallel and close to each other. The patient is asked to perform hip and lumbar flexion without bending the knees. The distance from the tip of the patient's 3rd finger to the ground is measured at the last point that can be reached. The hand-to-ground distance is accepted as 0 cm for women and 10 cm for men. If the patient has excessive hamstring muscle shortness, hamstring stretching will be performed before the test.
Schober Testi | Recorded 8 weeks and 3 months after the end of treatment
  In the Schober test, the patient stands with their feet 30 cm apart. The physiotherapist marks 5 cm below and 10 cm above the S2 vertebra level or the equivalent spina iliaca posterior superior (SIPS) level. The distance between these two points should be 15 cm. The patient is then asked to flex as much as possible and the distance between these points is measured again and subtracted from 15. This difference should be at least 5 cm. If the patient has excessive hamstring muscle shortness, hamstring stretching will be performed before the test.
Pain Catastrophizing Scale | Recorded 8 weeks and 3 months after the end of treatment
  The Pain Catastrophizing Scale is a self-report questionnaire used to examine pain catastrophizing. The scale consists of 13 statements that include a range of thoughts and feelings that an individual may experience when in pain. The items are divided into rumination, magnification, and helplessness categories, and each item is scored on a 5-point (0-4) scale.
Roland-Morris Disability Questionnaire | Recorded 8 weeks and 3 months after the end of treatment
  The Roland-Morris Disability Questionnaire is the most sensitive questionnaire for patients with mild to moderate disability due to acute, subacute or chronic low back pain. The patient is asked to mark a statement that applies to him/her on that day. The score ranges from 0 (no disability) to 24 (maximum disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moutzouri M, Perry J, Billis E. Investigation of the effects of a centrally applied lumbar sustained natural apophyseal glide mobilization on lower limb sympathetic nervous system activity in asymptomatic subjects. J Manipulative Physiol Ther. 2012 May;35(4):286-94. doi: 10.1016/j.jmpt.2012.04.016. PMID 22632588
- See also: Related Info — https://www.who.int/news-room/fact-sheets/detail/low-back-pain